CLINICAL TRIAL: NCT06178705
Title: Helpful Parenting Program (HPP) for Psychological Functioning of Parents of Children With Emotional and Behavioral Issues: A Randomized Control Trial
Brief Title: Parenting Program for Parents of Children With Emotional and Behavioral Issues: A Randomized Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Qasir Abbas, Dr. Qasir Abbas Assistant Professor Clinical Psychology, Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Govt.CUF
Record Dates: First submitted 2023-11-29; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Parent-Child Relations
Keywords: HPP, Parenting, Emotional & behavioral issues

STUDY DESIGN:
Intervention Model Description: Randomized control trial design would be used in this study which is two arm study having two groups, an experimental & wait-list control group. Experimental group will receive intervention while other group will be placed in wait-list. In this study, parallel group design would be used. The treatment will be given to all participants in a parallel way. Allocation ratio and framework would be equivalence i.e., equal number of participants in treatment and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Experimental Group:
  Participants in experimental group would receive 8-10 sessions of intervention based helpful parenting program
  Interventions: Behavioral: Helpful Parenting Program Intervention
- Control Group (No Intervention): Control Group:
  Participants in the control group will not receive the said intervention of helpful parenting program.

INTERVENTIONS:
Behavioral: Helpful Parenting Program Intervention — 8-10 sessions with 60 minutes duration once in a week will be conducted with the parents in group and one-on-one setting. Helpful parenting program would be based on social learning theory, behavior modification and couple counseling. The program will be used as an intervention strategy with parents to built insight about their child's emotional & behavioral issues. Different strategies to teach parenting skills will also be used as an intervention. Further more, this program will target parents' psychological distress and couples' problematic conflicts regarding parenting
  Arms: Treatment Group

SUMMARY:
The main objectives of the study are:

1. To find out the effectiveness of Helpful Parenting Program (HPP) for psychological functioning of children's parent having behavioral and emotional issues.
2. To decrease psychological distress among children's parent having behavioral and emotional issues.

DETAILED DESCRIPTION:
In this Helpful Parenting Program, N=200 participants would be enrolled for eligibility assessment from different schools in Faisalabad. 70 participants after the eligibility assessment and screening would be allocated to experimental and waitlist treatment condition. Participants would be allocated through random assignment using block randomization. In experimental group, the parents of children with emotional & behavioral issues will be included and 8 to 10 sessions of helpful parenting program would be provided to the parents. Each of the group will be comprised of n=35.

Eligibility Criteria:

Only parents with dysfunctional parenting practices, having children with emotional and behavioral issues would be a part of the study. Second, Only parents would be included in the study who score above 18 on SDQ-4. Only parents having children aged 5 to 12 years would be included in the study. Parents with major psychological disorders would be excluded from the study. The parent served as single parent would be excluded from the study.The participants would be taken from any socioeconomic status.

Interventions:

8-10 sessions with 60 minutes duration once in a week will be conducted with the parents in group and one-on-one setting. Helpful parenting program would be based on social learning theory, behavior modification and couple counseling. The program will be used as an intervention strategy with parents to built insight about their child's emotional & behavioral issues. Different strategies to teach parenting skills will also be used as an intervention. Further more, this program will target parents' psychological distress and couples' problematic conflicts regarding parenting.

Expected Outcomes:

This study will help to provide valuable information to mental health professionals to understand and develop guidelines for parents of children with emotional & behavioral issues. Further, this program would decrease psychological distress & couple's problematic conflicts among parents and improve the psychological functioning of parents. Moreover, this program will improve parental competence and make them independent problem solvers.

ELIGIBILITY:
Inclusion Criteria:

* Only parents with dysfunctional parenting practices, having children with emotional and behavioral issues would be a part of the study. Second, Only parents would be included in the study who score above 18 on SDQ-4. Only parents having children aged 5 to 12 years would be included in the study. The participants would be taken from any socioeconomic status.

Exclusion Criteria:

* Parents with major psychological disorders would be excluded from the study. The parent served as single parent would be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Strength and difficulty questionnaire | 4 months
  This scale will assess the parents strength and difficulty dealing the child
Depression Anxiety and Stress Scale | 4 months
  This scale will assess the level of depression, anxiety and stress among the parents of emotionally disturbed child
Dyadic Adjustment Scale | 4 months
  This scale will assess the parents level of adjustment

SECONDARY OUTCOMES:
Parenting Scale | 4 months
  This scale will assess the level of parenting
Parents sense of competence scale | 4 months
  This scale will assess the sense of competence

CONTACTS AND LOCATIONS:
Overall Officials: Qasir Abbas, PHD, Principal Investigator — Government College University Faisalabad
Locations (1):
- Qasir Abbas, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No